CLINICAL TRIAL: NCT00034853
Title: A 12 Week Double-blind Randomized Trial, With a 12 Week Open-label Extension, to Investigate the Efficacy and Safety of Meloxicam Oral Suspension Administered Once Daily and Naproxen Oral Suspension Administered Twice Daily in Children With Juvenile Rheumatoid Arthritis
Brief Title: Meloxicam [Mobic] in Juvenile Rheumatoid Arthritis (JRA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 107.235; NCT00274482 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Arthritis, Juvenile Rheumatoid
MeSH Terms: conditions — Arthritis, Juvenile

INTERVENTIONS:
Drug: meloxicam oral suspension
Drug: naproxen oral suspension

SUMMARY:
To obtain safety, efficacy, pharmacokinetic and dosing information for meloxicam oral suspension in children with Juvenile Rheumatoid Arthritis (JRA)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of juvenile idiopathic arthritis (JIA) by International League of Associations for Rheumatology (ILAR) criteria; pauciarthritic, extended pauciarthritic, or polyarthritic current course of disease;
* active arthritis of at least 2 joints
* at least 2 other abnormal variables of the 5 remaining core set parameters
* require nonsteroidal anti-inflammatory drugs (NSAIDs)
* children aged 2-17 years

Exclusion Criteria:

* systemic course of juvenile idiopathic arthritis
* all rheumatic conditions not included in inclusion criteria; any clinical finding or abnormal clinically relevant lab (not due to JIA) that could interfere with conduct of clinical trial
* weight of 9 kg or less
* pregnancy or breast feeding
* females of childbearing potential who are sexually active and not using adequate contraception for at least 3 mos prior to and for duration of study
* history of bleeding disorder, gastrointestinal bleeding, or cerebrovascular bleeding
* peptic ulcer past 6 months
* more than 1 disease modifying anti-rheumatic drug (DMARD) or change in DMARD during 3 months prior
* change corticosteroids during 1 month prior
* systemic corticosteroids greater than 10 mg/d, hydroxychloroquine greater than 10/mg/d, cyclosporine greater than 5 mg/kg/d., methotrexate greater than 15 mg/m2/wk, cytotoxic agents, gold, D-penicilamine, sulfasalazine, glucosamine, and investigational products
* etanercept during 1 month prior; infliximab during 2 months prior; intra-articular corticosteroids during 1 month prior
* patients requiring concomitant other NSAID including topical (excluding ophthalmic)
* requirement for use of other NSAIDs, anticoagulants, phenothiazine, lithium, or ACTH
* insufficient effect or intolerability to naproxen or meloxicam
* known or suspected hypersensitivity to trial meds or their excipients
* requirement of chronic H2 antagonist
* history of asthma, nasal polyps, angioneurotic edema, or urticaria with aspirin or NSAIDs
* planned surgical procedures during study
* investigational drug exposure during this trial or within 30 days (or 6 half lives, whichever greater) prior
* previous participation in this trial
* patients with known drug or alcohol abuse
* patient, parent or legal representative unable to understand and to comply with protocol

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2000-12; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Responder rate by core set of outcome criteria (Juvenile Rheumatoid Arthritis Pediatric 30): global assessment disease activity; functional disability, number joints arthritis, limited motion; erythrocyte sedimentation rate; | week 12

SECONDARY OUTCOMES:
Individual core set outcome criteria; final global assessment of efficacy; tolerability; AE incidence and intensity; withdrawals; acetaminophen consumption; safety labs: physical examination; hospitalization for gastrointestinal (GI) SAE, GI AE | weeks 4, 8, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (37):
- United States (29):
  - 107.235.23 Arkansas Children's Hospital, Little Rock, Arkansas
  - 107.235.17 Valley Children's Hospital, Madera, California
  - 107.235.37, San Diego, California
  - 107.235.4 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 107.235.12 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 107.235.13 Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - 107.235.36 Arthritis Associates Clinical Research of South Florida, Delray Beach, Florida
  - 107.235.21 Miami Children's Hospital, Miami, Florida
  - 107.235.38 Clinical Research Dept #7006, Saint Petersberg, Florida
  - 107.235.8 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 107.235.7 Boehringer Ingelheim Investigational Site, Kansas City, Kansas
  - 107.235.25 University of Louisville, Louisville, Kentucky
  - 107.235.16 Children's Hospital - Department of Rheumatology, New Orleans, Louisiana
  - 107.235.26 Deparment of Rheumatology, Boston, Massachusetts
  - 107.235.2 E15 Mayo Clinic, Rochester, Minnesota
  - 107.235.18 Washington University School of Medicine, St Louis, Missouri
  - 107.235.9 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 107.235.31 Department of Pediatrics, Omaha, Nebraska
  - 107.235.35 Arthritis and Rheumatic Disease Center, Livingston, New Jersey
  - 107.235.24 The Children's Hospital of Buffalo, Buffalo, New York
  - 107.235.19 Columbia Presbyterian Medical Center, New York, New York
  - 107.235.22 Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - 107.235.33 Healthcare Research Consultants, Tulsa, Oklahoma
  - 107.235.32 Arthritis and Osteoporosis Center, Duncansville, Pennsylvania
  - 107.235.39 Division of Ambulatory Pediatrics, Providence, Rhode Island
  - 107.235.10 Texas Scottish Rite Hospital, Dallas, Texas
  - 107.235.1 University of Utah School of Medicine, Salt Lake City, Utah
  - 107.235.30 Children's Hospital, Seattle, Washington
  - 107.235.20 Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (3):
  - 107.235.61, Cerqueira César
  - 107.235.62, Santa Cecília
  - 107.235.60, São Paulo
- 107.235.40, México, D.F., Mexico
- Ukraine (4):
  - 107.235.71 Institute of Children and Adolescents Health, Kharkiv
  - 107.235.70 Children Clinical Hospital No. 1, Kiev
  - 107.235.72 Institute of Pediatrics, Kiev
  - 107.235.73 2nd Children Specialized Clinical Hospital "OHMADIT", Kiev